CLINICAL TRIAL: NCT05439265
Title: Effect of an Electronic Medical Record Tool on the Documentation and Management of Newly Suspected Heparin Induced Thrombocytopenia
Brief Title: EMR Tool Impact on HIT Documentation and Management
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16092401-IRB01
Record Dates: First submitted 2016-10-18; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Heparin; Thrombocytopenia; Electronic Health Records
Keywords: HIT; Heparin Induced Thrombocytopenia; Electronic Medical Record; Electronic Health Records
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prior to 11/01/2014: Group prior to the implementation of an electronic medical record order panel and pharmacy resident involvement
- After 11/30/2014: Group after implementation of an electronic medical record order panel and pharmacy resident involvement
  Interventions: Other: Electronic medical record order panel and resident involvement

INTERVENTIONS:
Other: Electronic medical record order panel and resident involvement — Prior to 2014, there was no formal process for evaluation of patients with HIT. In November of 2014, an EMR tool was created in an effort to improve heparin allergy documentation and HIT management. This EMR tool prompts the medical team to perform the 4T score, displays the appropriate HIT labs, alternative anticoagulation strategies, instructs the nurse to apply an allergy bracelet, and notifies the pharmacy resident through the order verification queue. The pharmacy resident then performs an independent 4T score, discontinues all heparin products, documents the heparin allergy in the medical record, and assesses the need for alternative anticoagulation.
  Groups: After 11/30/2014

SUMMARY:
Heparin-induced thrombocytopenia (HIT) is an immune-mediated adverse drug reaction to heparin products which results in a prothrombotic state. Heparin-induced thrombocytopenia generally occurs several days after the start of unfractionated heparin or low molecular weight heparin and is diagnosed based on clinical presentation, and presence of thrombocytopenia. HIT has an incidence of 0.1% to 5% and if recognized early can help prevent major complications. As of November 2014, the responsibility for documenting heparin allergies in the electronic medical record (EMR) has shifted from the physician/medical resident to the pharmacy resident. The purpose of this study is to compare the number, rate, and appropriateness of heparin allergy documentation in order to help decrease adverse medical events related to heparin.

DETAILED DESCRIPTION:
Heparin-induced thrombocytopenia is a unique form of drug induced thrombocytopenia associated with increased clotting risk. The incidence of HIT ranges from 0.1% to 5%. Heparin-induced thrombocytopenia occurs when an antibody forms a complex with platelet factor 4 and heparin. This complex activates platelets which increases the risk of thrombus formation. Normally, HIT presents 5 to 14 days after exposure, but can occur with heparin exposure within the past 100 days. The presentation of HIT is often first suspected secondary to a decrease in platelet counts of 50% or more from baseline.

At Rush University Medical Center (RUMC), HIT is diagnosed through a combination of clinical factors and laboratory tests. When HIT is first suspected, a 4T HIT score, which is used to estimate the probability of true HIT, is calculated. The following score ranges correspond to the probability of true HIT; score of 0-3 indicates a low probability, score of 4-5 indicates an intermediate probability, and a score of 6-8 indicates a high probability of true HIT.

If the score indicates a likelihood of HIT, a HIT-Ab is sent off. This test has a sensitivity of more than 95% and a specificity of 74% to 86%. Accordingly, if this HIT-Ab test result is negative, HIT is ruled out. If the result is equivocal or positive, a confirmatory Serotonin Release Assay (SRA) test should be performed (sensitivity of 89% to 100% and a specificity of 88 % to 100%).

Prior to 2014, there was no formal process for evaluation of patients with HIT. In November of 2014, an EMR tool was created in an effort to improve heparin allergy documentation and HIT management. This EMR tool prompts the medical team to perform the 4T score, displays the appropriate HIT labs, alternative anticoagulation strategies, instructs the nurse to apply an allergy bracelet, and notifies the pharmacy resident through the order verification queue. The pharmacy resident then performs an independent 4T score, discontinues all heparin products, documents the heparin allergy in the medical record, and assesses the need for alternative anticoagulation.

Many studies have shown the value of the 4T HIT scoring system and the use of pharmacists in reducing the inappropriate use of alternative anticoagulation and unnecessary testing. Pharmacists have helped to improve patient outcomes and decrease costs associated with HIT. The purpose of this study is to evaluate the impact of an EMR tool and pharmacy residents on allergy documentation and the management of HIT.

ELIGIBILITY:
Inclusion Criteria:

* HIT-Ab ordered
* Aged ≥ 18 years of age

Exclusion Criteria:

* Previously documented and confirmed HIT allergy prior to placement for new HIT-Ab
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be retrospective, and collected data will be a result of routine care. Adult patients 18 years of age or older with an order for a HIT-Ab while admitted to RUMC will be assessed for inclusion
  Patients will be reviewed from 01/01/2014 to 09/30/2015. A list of patients will be generated by a laboratory order for HIT-Ab (Heparin Induced Thrombocytopenia AB [LAB0002639]).
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2014-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Assess appropriate allergy documentation | From the date of first ordering of a HIT-Ab until HIT allergy is determined as positive or negative, assessed up to 4 weeks
  1. Completion of appropriate allergy documentation will include all of the following:
  a. Heparin allergy documented i. Pending result ii. Positive result b. Heparin allergy removed i. Negative result

SECONDARY OUTCOMES:
Administration of heparin products with pending HIT-Ab | From the date of first ordering of a HIT-Ab until HIT allergy is determined as positive or negative, assessed up to 4 weeks
  a. Defined as ordering of HIT-Ab or 4T score greater than 5 i. Low Probability: 0-3 ii. Intermediate Probability: 4-5 iii. High Probability: 6-8
Documentation of 4T HIT score in patient medical record | From the date of first ordering of a HIT-Ab until HIT allergy is determined as positive or negative, assessed up to 4 weeks
  Defined as documentation in a patient medical note, i-vent, or lab result
Initiation or withholding of Direct Thrombin Inhibitor (DTI) appropriate based on probability of HIT as scored by the 4T HIT score | From the date of first ordering of a HIT-Ab until HIT allergy is determined as positive or negative, assessed up to 4 weeks
  1. Initiation appropriate for 4T HIT score of greater than 5
  2. Withholding appropriate for 4T HIT score of 3 or less (in absence of clot)
Number of Serotonin Release Assay labs drawn appropriately | From the date of first ordering of a HIT-Ab until HIT allergy is determined as positive or negative, assessed up to 4 weeks
  1. Appropriate defined as drawn secondary to a positive HIT-Ab
  2. Inappropriate defined as drawn prior to ordering a HIT-Ab
Positive and negative predictive value of 4T score when performed by medical resident | From the date of first ordering of a HIT-Ab until HIT allergy is determined as positive or negative, assessed up to 4 weeks
  1. The percent of all positive tests that are true positives is the Positive Predictive Value.
  2. The percent of all negative tests that are true negatives is the Negative Predictive Value
Positive and negative predictive value of 4T score when performed by pharmacy residents | From the date of first ordering of a HIT-Ab until HIT allergy is determined as positive or negative, assessed up to 4 weeks
  1. The percent of all positive tests that are true positives is the Positive Predictive Value.
  2. The percent of all negative tests that are true negatives is the Negative Predictive Value

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Peksa, PharmD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kniuksta, Ruth, Amy Mozina, and Peggy Reed.
- [Background] Konkle B. Chapter 115. Disorders of Platelets and Vessel Wall. In: Longo DL, Fauci AS, Kasper DL, Hauser SL, Jameson J, Loscalzo J. eds. Harrison's Principles of Internal Medicine, 18e. New York, NY: McGraw-Hill; 2012. Accessed August 14, 2016.
- [Result] Hasan M, Malalur P, Agastya M, Malik AO, Dawod Y, Jaradat M, Yoo JW, Makar R. A high-value cost conscious approach to minimize heparin induced thrombocytopenia antibody (HITAb) testing using the 4T score. J Thromb Thrombolysis. 2016 Oct;42(3):441-6. doi: 10.1007/s11239-016-1396-6. PMID 27377975
- [Result] Bayat M, Macedo FY, Ansari AS, Bracey AW, Akinyele S, Salazar M. Evaluation of clinical and laboratory data for early diagnosis of heparin-induced thrombocytopenia. Am J Health Syst Pharm. 2015 Oct 1;72(19):1649-55. doi: 10.2146/ajhp140778. PMID 26386106
- [Result] Andreescu AC, Possidente C, Hsieh M, Cushman M. Evaluation of a pharmacy-based surveillance program for heparin-induced thrombocytopenia. Pharmacotherapy. 2000 Aug;20(8):974-80. doi: 10.1592/phco.20.11.974.35264. PMID 10939559
- [Result] Smythe MA, Mehta TP, Koerber JM, Forsyth LL, Sykes E, Corbets LR, Melendy SM, Parikh R. Development and implementation of a comprehensive heparin-induced thrombocytopenia recognition and management protocol. Am J Health Syst Pharm. 2012 Feb 1;69(3):241-8. doi: 10.2146/ajhp110313. PMID 22261947
- [Result] Burnett AE, Bowles H, Borrego ME, Montoya TN, Garcia DA, Mahan C. Heparin-induced thrombocytopenia: reducing misdiagnosis via collaboration between an inpatient anticoagulation pharmacy service and hospital reference laboratory. J Thromb Thrombolysis. 2016 Nov;42(4):471-8. doi: 10.1007/s11239-016-1381-0. PMID 27229333
- [Result] Floresca D, Dupree L, Basile S, Tan P. Evaluation of appropriate serologic testing for suspected heparin-induced thrombocytopenia. Am J Health Syst Pharm. 2012 Sep 15;69(18):1581-7. doi: 10.2146/ajhp110513. PMID 22935941